CLINICAL TRIAL: NCT07125755
Title: A Prospective, Multicenter, Randomized Controlled Phase 3 Clinical Trial Comparing Postoperative Adjuvant Cisplatin Concurrent Chemoradiotherapy With Adjuvant Radiotherapy Alone for Intermediate-risk Head and Neck Squamous Cell Carcinoma
Brief Title: Comparing Postoperative Adjuvant Cisplatin Concurrent Chemoradiotherapy With Adjuvant Radiotherapy Alone for Intermediate-risk Head and Neck Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lei Chen, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SL-B2025-367-02
Record Dates: First submitted 2025-08-10; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Squamous Cell Cancer of Head and Neck (SCCHN)
Keywords: Concurrent chemoradiotherapy; Cisplatin; postoperative head and neck squamous cell carcinoma
MeSH Terms: interventions — Cisplatin

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2 courses of cisplatin chemoradiotherapy arm (Experimental): Patients will receive intensity modulated radiotherapy (total dose: > 66 Gy, split dose: 2-2.2 Gy/ time, once a day, 5 times a week) plus concurrent Cisplatin chemotherapy (100 mg/m2 intravenous injection,once every 3 weeks, twice in total, on days 1 and 22).
  Interventions: Drug: Cisplatin
- Postoperative adjuvant radiotherapy alone (No Intervention): Patients will receive intensity modulated radiotherapy (total dose: > 66 Gy, split dose: 2-2.2 Gy/ time, once a day, 5 times a week)

INTERVENTIONS:
Drug: Cisplatin — Concurrent Cisplatin chemotherapy (100 mg/m2 intravenous injection,once every 3 weeks, twice in total, on days 1 and 22) will be given plus intensity modulated radiotherapy
  Arms: 2 courses of cisplatin chemoradiotherapy arm

SUMMARY:
The main objective of this trial was to determine the value of concurrent chemoradiotherapy for Intermediate-risk head and neck squamous cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

A. The pathological type is head and neck squamous cell carcinoma

* Stages

B. Radical surgery has been performed, and there are intermediary-risk factors (pT3/pT4, pN2/pN3, positive lymph nodes in the cervical IV/V region of oral cancer, nerve invasion, and vascular invasion).

C. No evidence of distant metastasis (M0).

D. Functional status: Karnofsky scale (KPS) > 70.

E. Normal bone marrow function:

* white blood cell count > 4×109/L
* hemoglobin > 120g/L in males, 110g/L in females
* platelet count > 100×109/L

G. Normal liver function:

* alanine aminotransferase (ALT), aspartate aminotransferase (AST) < 1.5 times the upper limit of normal (ULN)
* alkaline phosphatase (ALP) < 2.5×ULN
* bilirubin < ULN.

H. Normal renal function: creatinine clearance > 60 ml/min.

I. Patients must be informed of the basic contents of this study and sign informed consent.

Exclusion Criteria:

A. Age >70 years or <18 years.

B. Treatment is palliative.

C. Previous chemotherapy (except induction chemotherapy prior to surgery).

D. Previous radiation therapy.

E. Women who are pregnant or breastfeeding

F. Previous history of malignant tumor.

G. With other serious medical conditions that may pose a greater risk or affect compliance with the test. Examples include:

* unstable heart disease that requires treatment
* kidney disease
* chronic hepatitis
* poorly controlled diabetes (fasting blood glucose > 1.5×ULN)
* mental illness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2028-08-15 (Estimated); Study Completion 2031-08-15 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival (FFS) | 3 years
  calculated from enrolment to the date of locoregional recurrence,distant metastasis,or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  calculated from enrolment to the date of death from any cause.
Distant metastasis-free survival(DMFS) | 3 years
  calculated from enrolment to the date of first distant metastasis.
locoregional recurrence-free survival (LRRFS) | 3 years
  calculated from enrolment to the date of locoregional persistence or 1st locoregional recurrence.
Quality of life (QoL) | 3 years
  The change of QoL from randomization to the start of radiotherapy,the end of radiotherapy,13-16 weeks after radiotherapy,2 years and 3 years after randomization. The EORTC QoL questionnaire-C30(EORTC quality of life questionnaire-C30#version 3.0 will be used. This questionnaire comprises 30 questions,24 of which are aggregated into nine multi- question scales,that is,five functioning scales (e.g.,physical),three symptom scales (e.g.,fatigue)and one global health status scale. The remaining six single-question (e.g.,dyspnoea)scales assess symptoms. These 15 scales will be scored according to the official Scoring Manual.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Chen Principal Investigator, M.D, Principal Investigator — Sun Yat-sen University
Locations (6):
- China (6):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Affiliated Hospital of Guilin Medical College, Guilin, Guangxi
  - Hainan General Hospital, Sanya, Hainan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No